CLINICAL TRIAL: NCT07090044
Title: Comparing Post-intravitreal Injection Pain Scores Using Loteprednol, Bromfenac Sodium, and Artificial Tears Over a 24-hour Period
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Retina Research Institute, LLC (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19928
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Vein Occlusion; Macular Degeneration Choroidal Neovascularization; Macular Edema; Diabetic Retinopathy
Keywords: Intravitreal Injection; Post-procedure Pain
MeSH Terms: conditions — Choroidal Neovascularization; Macular Edema; Diabetic Retinopathy | interventions — Loteprednol Etabonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bromfenac (Active Comparator): Bromfenac sodium 0.07% is a nonsteroidal anti-inflammatory drug to be administered as a topical drop in the eye receiving the standard of care intravitreal injection.
  Interventions: Drug: Bromfenac Sodium 0.07%
- Loteprednol (Active Comparator): Loteprednol etabonate ophthalmic gel 0.38% is a steroidal drug to be administered as a topical drop in the eye receiving the standard of care intravitreal injection.
  Interventions: Drug: Loteprednol Etabonate 0.38% Ophthalmic Gel/Jelly
- Artificial Tears (Placebo Comparator): Propylene Glycol Preservative-free artificial tears is a placebo comparator to be adminstered in the eye receiving the standard of care intravitreal injection.
  Interventions: Drug: Propylene Glycol Preservative-free Artificial Tears

INTERVENTIONS:
Drug: Bromfenac Sodium 0.07% — Bromfenac sodium 0.07% is a nonsteroidal anti-inflammatory drug to be administered as one topical drop, one time 5 minutes prior to the regularly scheduled standard of care intravitreal injection.
  Arms: Bromfenac
Drug: Loteprednol Etabonate 0.38% Ophthalmic Gel/Jelly — Loteprednol etabonate 0.38% ophthalmic gel is a steroidal drug to be administered as one topical drop three times daily on the day of the regularly scheduled standard of care intravitreal injection. The first drop administered 5 minutes prior to the intravitreal injection.
  Arms: Loteprednol
Drug: Propylene Glycol Preservative-free Artificial Tears — Propylene Glycol Preservative-free Artificial Tears is a placebo compartor administered as one topical drop three times daily on the day of the regularly scheduled standard of care intravitreal injection. The first drop administered 5 minutes prior to the intravitreal injection.
  Arms: Artificial Tears

SUMMARY:
The goal of this clinical trial is to learn how various topical drops (bromfenac, loteprednol, and artificial tears) fare in alleviating post-intravitreal injection pain. The main questions it aims to answer are:

- Do bromfenac sodium and/or loteprednol etabonate improve post-injection pain scores compared to preservative-free artificial tears?

Participants will:

* Receive one drop of the topical drops five minutes prior to their regularly scheduled intravitreal injection. Depending on the treatment arm, they will also administer drops on their own at home up to 3 times per day on the day of their procedure.
* They will answer a standardized pain score survey at 4 hours and 24 hours following their intravitreal injection and convey their results to study coordinators by phone.

ELIGIBILITY:
Inclusion Criteria:

* Standard of Care Treatment with intravitreal injection
* History of at least 1 anti-VEGF injection in the 90 days prior to inclusion
* Less than 13 intravitreal injection in the 365 days prior to inclusion

Exclusion Criteria:

* History of autoimmune disease, graft versus host disease, neurotrophic corneal disease, contact lens use, keratitis, fibromyalgia, uveitis, herpetic ocular disease
* Drug allergy to any drug components
* History of any ocular surgery in the 30 days prior to inclusion
* Current topical corticosteroid or non-steroidal anti-inflammatory drug (NSAID)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Pain Score | At 4 hours and 24 hours following intravitreal injection
  A standardized Visual Analog Scale (VAS) pain score is collected at 4 hours and 24 hours following standard of care intravitreal injection. Patients are provided a VAS scale and receive a call from study coordinators to collect pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sabin Dang, MD, Principal Investigator — Retina Research Institute, LLC
Locations (1):
- The Retina Institute, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD Collected throughout the trial
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] SakallioGlu AK, Kaya S, GarIp R, Guclu H. COMPARISON OF THE EFFECTS OF EIGHT DIFFERENT TOPICAL NONSTEROIDAL ANTI-INFLAMMATORY DRUGS ON REDUCING INTRAVITREAL INJECTION-INDUCED PAIN. Retina. 2024 Jul 1;44(7):1196-1202. doi: 10.1097/IAE.0000000000004085. PMID 38437826
- [Background] Lee DH, Kim M, Choi EY, Chin HS, Kim M. Efficacy of Pretreatment with Preservative-Free Topical Bromfenac in Improving Post-Intravitreal-Injection Pain: A Prospective Pilot Study. J Clin Med. 2022 Jul 18;11(14):4172. doi: 10.3390/jcm11144172. PMID 35887936
- [Background] Rifkin L, Schaal S. Shortening ocular pain duration following intravitreal injections. Eur J Ophthalmol. 2012 Nov-Dec;22(6):1008-12. doi: 10.5301/ejo.5000147. Epub 2012 Apr 24. PMID 22562296
- [Background] Shtayer C, Lily Okrent Smolar A, Elmalak M, Abayev L, Grzybowski A, Moisseiev E. Post-Intravitreal injection pain reduction using topical NSAIDS: A comparative study. Eur J Ophthalmol. 2025 Sep;35(5):1703-1709. doi: 10.1177/11206721231201176. Epub 2023 Sep 10. PMID 37691285
- [Background] Georgakopoulos CD, Tsapardoni F, Makri OE. EFFECT OF BROMFENAC ON PAIN RELATED TO INTRAVITREAL INJECTIONS: A Randomized Crossover Study. Retina. 2017 Feb;37(2):388-395. doi: 10.1097/IAE.0000000000001137. PMID 27442130
- [Background] Popovic MM, Muni RH, Nichani P, Kertes PJ. Topical Nonsteroidal Anti-inflammatory Drugs for Pain Resulting from Intravitreal Injections: A Meta-Analysis. Ophthalmol Retina. 2020 May;4(5):461-470. doi: 10.1016/j.oret.2020.01.024. Epub 2020 Feb 13. PMID 32199867